CLINICAL TRIAL: NCT04411394
Title: The Validity and Reliability Study of Turkish Version of Body Perception Questionnaire
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: Yeditepe.U
Record Dates: First submitted 2020-05-05; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Body Image
Keywords: Anxiety; Body Perception Questionnaire; Interoception; Validity; Reliability
MeSH Terms: conditions — Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Participants: There is no intervention
  Interventions: Other: Questionnaire
- Anxiety Participants: There is no intervention
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Body Perception Questionnaire and Hospitalized Anxiety and Depression Scale

SUMMARY:
The present study aims to determine the validity and reliability of the Turkish version of the Body Perception Questionnaire (BPQ) through the Turkish translation of the questionnaire and the intercultural adaptation. The Body Perception Questionnaire (BPQ) is a self-report measure of body awareness and autonomic reactivity. Its items are based on the organization of the autonomic nervous system (ANS), a set of neural pathways connecting the brain and body.

DETAILED DESCRIPTION:
The present study aims to determine the validity and reliability of the Turkish version of the "Body Perception Questionnaire (BPQ) through the Turkish translation of the questionnaire and the intercultural adaptation. The Body Perception Questionnaire (BPQ) is a self-report measure of body awareness and autonomic reactivity. Its items are based on the organization of the autonomic nervous system (ANS), a set of neural pathways connecting the brain and body. These pathways send information from the body about the status of organs and tissues (i.e., afferent projections). Some of these incoming signals form a basis for the subjective awareness of the body. The ANS also carries signals that control the functions of these organs and tissues (i.e., efferent projections). These signals can alter the functions of the body, depending on internal and external needs. The study includes 175 healthy participants and 120 participants with anxiety. Beaton's 6-step procedure was used for translation and intercultural adaptation. After the steps of the procedure were completed, the questionnaire was finalized.

ELIGIBILITY:
Inclusion Criteria:

* Being a volunteer to participate in the study
* Being between the age of 18 - 77
* Understand and follow commands
* Not diagnosed a psychiatric disorder

Exclusion Criteria:

* Younger than the age of 18
* Reported taking psychotropic drugs and/or beta-blockers
* Did not complete the questions
* Having any surgical operation in the last six months
* Diagnosed chronic cardiovascular, pulmonary or neuromuscular systemic disorder

Ages: 18 Years to 77 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Marmara Region
Sampling Method: Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Body Perception Questionnaire | through study completion, an average of 1 year
  To understand the body perception
Hospitalized Anxiety and Depression Scale | through study completion, an average of 1 year
  To understand if they have anxiety problem

CONTACTS AND LOCATIONS:
Overall Officials: Feryal Subaşı, Professor, Study Chair — Yeditepe University, Faculty of Health Science; Aymen Balıkçı, MD, Study Chair — Sense On
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)